CLINICAL TRIAL: NCT01525459
Title: Monitoring and Analysis of Gene Expression, Immunological Status and Metabolome in Peripheral Blood Mononuclear Cells and Their Specific Subpopulations (CD4+ T Cells and CD56+ NK Cells) in Surgically Treated Glioma Patients
Brief Title: Gene Expression, Immunological Status and Metabolome in Glioma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Biology, Slovenia (Other Government)
Collaborators: Blood Transfusion Centre of Slovenia (Other Government); University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Tamara Lah Turnsek, Director of the National Institute of Biology, Slovenia, National Institute of Biology, Slovenia
Other Study IDs: MNC-Glioma-1-4
Record Dates: First submitted 2012-01-20; First posted 2012-02-03 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Glioma
Keywords: Glioma; PBMC subpopulations; Gene expression; Metabolomics; Immunological status; miRNA; Proteomics
MeSH Terms: conditions — Glioma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, blood plasma, peripheral blood mononuclear cells, CD4+ T cells, CD56+ NK cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glioma patients
  Interventions: Procedure: Glioma resection; Other: Blood sampling

INTERVENTIONS:
Procedure: Glioma resection — Patients will be treated with the standard surgical therapy - glioma resection.
Other: Blood sampling — Blood samples used for measuring studied parameters will be taken within 10 days before surgery, one day after surgery and once more within 10 days following the operative procedure.

SUMMARY:
Study on glioma patients treated with brain surgery is focusing on the analysis of their transcriptome expression profile measured in two immune cell populations, CD4+ T cells and CD56+ NK cells. The results of analysis will be compared to the reference data of healthy population. Furthermore, the metabolomic and immunological status will also be monitored and compared to healthy group reference data, before and after the surgery*. With comparative crossomics analysis the investigators intend to possibly identify new diagnostic and prognostic biological markers for the relapse of the disease. The results are expected to convey a deeper insight into pathophysiology of the glioma as well as into the mechanisms of the current surgical therapy.

* The healthy reference data have been published in collaborative efforts of BTC, UMC and NIB (Gruden et al. 2012).

ELIGIBILITY:
Inclusion Criteria:

* malignant glioma = glioblastoma (WHO IV) patients

Exclusion Criteria:

* pregnancy
* metastases

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glioma patients treated with surgical resection of the tumor
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Transcriptome profile of CD4+ T and CD56+ NK cells | within 10 days before surgery
Transcriptome profile of CD4+ T and CD56+ NK cells | one day after surgery
Transcriptome profile of CD4+ T and CD56+ NK cells | within 10 days after surgery

SECONDARY OUTCOMES:
Metabolite profiling in blood plasma samples | within 10 days before surgery, one day after surgery and once more within 10 days after surgery surgery
Lymphocyte subpopulation assessment in peripheral blood samples | within 10 days before surgery, one day after surgery and once more within 10 days after surgery
Antibody profiling in blood plasma samples | within 10 days before surgery, one day after surgery and once more within 10 days after surgery
miRNA profiling in blood plasma samples | within 10 days before surgery, one day after surgery and once more within 10 days after surgery surgery
Proteomic analysis of blood plasma samples | within 10 days before surgery, one day after surgery and once more within 10 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Lah Turnšek, PhD, Study Chair — National Institute of Biology, Ljubljana, Slovenia; Kristina Gruden, PhD, Principal Investigator — National Institute of Biology, Ljubljana, Slovenia
Locations (3):
- Slovenia (3):
  - Blood Transfusion Centre of Slovenia, Ljubljana
  - Department of Neurosurgery, University Medical Centre Ljubljana, Ljubljana
  - National Institute of Biology, Ljubljana

REFERENCES:
- [Background] Gruden K, Hren M, Herman A, Blejec A, Albrecht T, Selbig J, Bauer C, Schuchardt J, Or-Guil M, Zupancic K, Svajger U, Stabuc B, Ihan A, Kopitar AN, Ravnikar M, Knezevic M, Rozman P, Jeras M. A "crossomics" study analysing variability of different components in peripheral blood of healthy caucasoid individuals. PLoS One. 2012;7(1):e28761. doi: 10.1371/journal.pone.0028761. Epub 2012 Jan 12. PMID 22253695
- See also: Official internet page of the Slovenian National Institute of Biology — http://www.nib.si
- See also: Official internet page of the project SYSTHER (Systems Biology Tools Development For Cell Therapy And Drug Development) — http://systher.biologie.hu-berlin.de